CLINICAL TRIAL: NCT01031017
Title: Prophylactic Administration of Natural Progesterone in the Prevention of Preterm Delivery in Twin Pregnancies: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Prophylactic Administration of Natural Progesterone in the Prevention of Preterm Delivery in Twin Pregnancies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Maria de Lourdes Brizot, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 418/04
Record Dates: First submitted 2009-12-09; First posted 2009-12-14 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Preterm Delivery
Keywords: twin pregnancies; preterm delivery; progesterone
MeSH Terms: conditions — Premature Birth | interventions — Progesterone; Utrogestan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): group taking placebo
  Interventions: Drug: placebo
- study group (Active Comparator): group taking progesterone
  Interventions: Drug: progesterone

INTERVENTIONS:
Drug: progesterone — ovules, 200mg per vagina, once a day from 18 weeks
  Other Names: utrogestan
  Arms: study group
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
Twin pregnancies are at substantial increased risk of preterm delivery. Prophylactic administration of progesterone in singleton pregnancies at risk of preterm delivery has been shown to be effective in reducing the rate of such complication. The aim of this study is to investigate the effect of prophylactic administration of natural progesterone in twin pregnancies on the rate of preterm births.

DETAILED DESCRIPTION:
In a double-blind, placebo controlled study performed in our Institution, Fonseca et al., investigated the use of micronized natural progesterone, crafted in vaginal capsules of 100mg, for the prevention of preterm delivery. The study involved 142 singleton pregnancies at high risk for premature birth (previous premature birth, cerclage and uterine malformation). The progesterone was introduced from 24 weeks to 34 weeks gestation. The authors observed a significant reduction of premature birth before 37 weeks (28,1% within the placebo group versus 13,8% within the treated group) and below 34 weeks (18,6% within the placebo group versus 2,8% within the treated group). Also, it was observed a reduction in the frequency of the uterine contractions in the progesterone group.

In the only study performed specifically among twin pregnancies, Anna Lisa et al. in 1980, administrated 250mg of 17αOH-PC or placebo (still oil) weekly, in 70 pregnant women with twin pregnancies, beginning before 28 weeks and continuing up to 37 weeks gestation. Seric levels of progesterone, estradiol, estriol, testosterone, and placental lactogenic hormone were also measured weekly. The differences among the achieved results within both groups, according the average in pregnancy duration (36,9 within the treated group, versus 37,3 within the placebo group), the average birthweight and the perimortality rate were not significantly different, as well as the levels of progesterone, estriol, estradiol, testosterone and placental lactogenic hormone. Nevertheless, this study was criticized for starting the use of progesterone at a late stage of pregnancy, in a considerable number of cases.

These studies suggest that in singleton pregnancies with a previous history of preterm birth progesterone treatment may prevent the patients from having subsequent premature births. Nonetheless, the results of these series must not be generalized to all pregnancies at high risk. Additional studies to evaluate the use of progesterone ovules in multiple pregnancies are necessary, as these pregnancies are increasing due to the advanced maternal age at the conception time and also due to the widespread use of assisted reproductive techniques.

ELIGIBILITY:
Inclusion Criteria:

* Naturally conceived diamniotic twin pregnancies.
* Absence of major fetal abnormalities (such as neural tube defects, abdominal wall defects, cardiac defects, hydrocephalus, malformations that course with polyhydramnios) at the anomaly scan.
* Gestational age between 18 - 21+6weeks at the moment of randomization.
* Patients that are not allergic to the progesterone capsule excipients (arachis oil, soy and lecithin).
* Patients who do not use other medicines that can alter the progesterone effects, such as: barbituric, carbamazepine, hydantoin, rifampicin, betablockers, teofiline or ciclosporin.
* Porphyria, otoscleroses, malignant disease or severe depressive state.

Exclusion Criteria:

* Premature rupture of membranes diagnosed at the moment of recruitment.
* Subsequent diagnosis of major fetal abnormalities.
* Twin to twin transfusion syndrome diagnosed during the course of the pregnancy.
* Presence of ovular infection.
* Death of one or both fetuses in any time of the pregnancy.
* Giving up or discontinuing the use of the medication.
* Elective or iatrogenic premature birth (before 34 weeks).
* Present or past history of thromboembolic disease
* Uterine malformation
* Known or suspected breast or genitals malignancy tumor
* Plan to move to another city during pregnancy
* Placenta Previa

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 390 (Actual)
Dates: Start 2007-06; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
gestational age at delivery | once at the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Maria Brizot, PhD, Principal Investigator — Department of Obstetrics, São Paulo University Medical School
Locations (1):
- Hospital das Clinicas, São Paulo, São Paulo, Brazil